CLINICAL TRIAL: NCT01191320
Title: A Study to Evaluate the Efficacy of Androxal® in Improving Glycemic Control in Men With Secondary Hypogonadism or Adult-onset Idiopathic Hypogonadotropic Hypogonadism (AIHH) and Type 2 Diabetes Mellitus With Sub-Optimum Treatment
Brief Title: Study to Evaluate the Efficacy of Androxal in Controlling Blood Glucose in Men With Type-2 Diabetes Mellitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Repros Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZA-202
Record Dates: First submitted 2010-08-27; First posted 2010-08-30 (Estimated); Results first posted 2014-07-24 (Estimated); Last update posted 2014-07-24 (Estimated); Status verified 2014-06

CONDITIONS: Type 2 Diabetes Mellitus; Secondary Hypogonadism
Keywords: Adult onset hypogonadotropic hypogonadism
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypogonadism | interventions — Enclomiphene

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- Androxal 12.5 mg (Experimental): 12.5 mg/day
  Interventions: Drug: Androxal
- Androxal 25 mg (Experimental): 25 mg/day
  Interventions: Drug: Androxal

INTERVENTIONS:
Drug: Placebo — Placebo capsule 1x daily for 3 months
  Arms: Placebo
Drug: Androxal — Capsules 12.5 mg or 25 mg 1x daily for 3 months
  Other Names: Enclomiphene citrate
  Arms: Androxal 12.5 mg; Androxal 25 mg

SUMMARY:
The purpose of this study is to determine the effect the investigative drug has on glycemic control in men with type 2 diabetes mellitus (T2DM) and secondary hypogonadism

DETAILED DESCRIPTION:
A phase IIB, multi-center, randomized, parallel, placebo- and active-controlled trial in adult male subjects with secondary hypogonadism who have been treated with OHAs but are not in glycemic control. All subjects currently treated with exogenous testosterone will discontinue at screening for at least 21 days and remain off testosterone for the course of the study. One hundred twenty to 150 subjects will be randomly assigned to one of three treatment groups according to a 1:1:1 ratio. Subjects will receive one of two dose strengths of Androxal or placebo in addition to their usual dose of mono- or combination OHAs for three months. Following an initial screening period, subjects will return monthly for 3 months and 1 month later for a follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Males, ages 20 to 80-years-old, inclusive
* A diagnosis of type 2 diabetes mellitus by American Diabetes Association (ADA) criteria for at least 6 months
* Treatment with a stable but sub-optimum dose of OHAs for at least 2 months prior to screening based on a lack of control of blood glucose
* Previous diagnosis of adult-onset idiopathic hypogonadotropic hypogonadism (AIHH) and have undergone treatment with a topical testosterone gel, Low-to-borderline morning total testosterone (TT), after at least a two week wash-out period, and normal or low normal serum luteinizing hormone (LH)at screening and at baseline
* No previous diagnosis of AIHH but present as naïve patients with low morning TT and normal or low normal serum LH at screening and at baseline
* Body Mass Index (BMI) between 26 and 40 kg/m2
* Fasting blood (plasma or serum) glucose (FBG) between 125 and 240 mg/dL
* HemoglobinA1c in serum as (HbA1c) between 7% and 9.5%
* Comprehends informed consent
* Otherwise normal healthy males
* All clinical laboratory test within normal ranges (any deviation outside the normal range will require approval of investigator)
* Ability to complete the study in compliance with the protocol
* Ability to understand and provide written informed consent

Exclusion Criteria:

* A history of testicular failure, Kallmann Syndrome or other infertility condition
* Clinically significant medical condition rendering the subjects infertile including tumors of the pituitary, laboratory abnormalities, or having received an investigational drug in the past 30 days prior to study
* Prostate nodules or induration, a history of, known, or suspect prostate cancer not ruled out by a negative biopsy, or a prostate specific antigen (PSA) higher than 3.5;
* Hematocrit in excess of 47% or a hemoglobin (Hb) greater than 16 g/dl
* Previous treatment with androgens, estrogens, DHEA, testosterone or testosterone analogues in injectable, oral, topical or other forms for the treatment of AIHH who have not discontinued at the start of the treatment phase;
* Primary hypogonadism as typified as a serum LH greater than 15 and a TT value less than 300 ng/dL
* Continuous use of corticosteroids
* History of or current diagnosis of major macrovascular complications of T2DM: myocardial infarction (MI) or stroke within 6 months, or any history of coronary revascularization, unstable angina, congestive heart failure (CHF) of New York Heart Association (NYHA) greater than or equal to 2
* Uncontrolled sitting blood pressure (BP) greater than 150/95, serum creatinine (Cr) greater than 1.5 ULN or estimated glomerular filtration rate (eGFR) less than mL/min/1.73 m2
* Retinopathy requiring continuing ophthalmologic assessments
* Cataracts
* Other significant history of diabetic complications (proteinuria greater than 1 g/d, retinopathy, clear neuropathy)
* Aspartate transaminase (AST), alanine transaminase (ALT), or alkaline phosphatase greater than 3 times the upper limits of normal (ULN)
* Total bilirubin greater than 2.0 mg/dL (>34 µmol/L);
* Injectable testosterone within 120 days of Screening (Visit 1)
* Reported substance abuse at screening
* Taking insulin therapy;
* Clinically significant abnormal findings on screening examination as determined by the investigator
* Known hypersensitivity to clomiphene citrate;
* Current or history of breast cancer
* Any condition which in the opinion of the investigator would interfere with the participant's ability to provide informed consent, comply with the study instructions, possibly confound interpretation of the study results, or endanger the participant if he took part in the study.

Ages: 20 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2010-10; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Cunningham, MD, Principal Investigator — Baylor College of Medicine
Locations (17):
- United States (17):
  - Paradigm Clinical Research, Garden Grove, California
  - Northern California Research Corp, Sacramento, California
  - LABioMed, Torrance, California
  - Lahey Clinic, Peabody, Massachusetts
  - Affiliated Clinical Research, Las Vegas, Nevada
  - Dr. Bruce Gilbert, Great Neck, New York
  - University Urology, New York, New York
  - Mount Sinai School of Medicine, New York, New York
  - Dr. Michael Werner, Purchase, New York
  - Discovery Clinical Trials, Austin, Texas
  - Research Across America, Carrollton, Texas
  - TX Urology Associate, Houston, Texas
  - Centex Research, Houston, Texas
  - Dr. Rakesh Patel, Houston, Texas
  - Protenium Clinical Research, Hurst, Texas
  - R/D Clinical Research, Lake Jackson, Texas
  - Cetero Research, San Antonio, Texas

REFERENCES:
- See also: Sponsor website — http://www.reprosrx.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Androxal 12.5 mg | Androxal 25 mg
Started | 43 | 38 | 38
Completed | 36 | 32 | 31
Not Completed | 7 | 6 | 7

BASELINE CHARACTERISTICS:
Population: Safety population
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Androxal 12.5 mg | Androxal 25 mg | Total
Number analyzed (Participants) | 43 | 38 | 38 | 119
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.3 (8.4) | 55.9 (9.5) | 57.6 (8.4) | 57.0 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 43 | 38 | 38 | 119
Region of Enrollment [Number; unit: participants]
  United States | 43 | 38 | 38 | 119
HgbA1c ratio [Mean (Standard Deviation); unit: Ratio] | 0.08 (0.012) | 0.08 (0.013) | 0.09 (0.017) | 0.08 (0.014)

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1C
Description: The change in HbA1c from Baseline to 3 Months for each treatment arm
Time Frame: 3 months
Population: ITT population
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Placebo | Androxal 12.5 mg | Androxal 25 mg
Number analyzed (Participants) | 43 | 38 | 35
Ratio | 0 (0.012) | 0 (0.015) | 0 (0.010)

ADVERSE EVENTS:
Arm/Group | Placebo | Androxal 12.5 mg | Androxal 25 mg
Serious Adverse Events (participants affected / at risk) | 1/43 | 0/38 | 1/38
Other Adverse Events (participants affected / at risk) | 1/43 | 8/38 | 5/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=43) | Androxal 12.5 mg (N=38) | Androxal 25 mg (N=38)
Coronary bypass (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) — Subject was hospitalized for triple bypass surgery considered by PI to be unrelated to treatment.
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) — Subject was hospitalized for severe chest pain. Study drug was continued. PI assessed as not related.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=43) | Androxal 12.5 mg (N=38) | Androxal 25 mg (N=38)
Sinusitis (Infections and infestations) | 0 | 2 | 1
Glycosylated Hemoglobin increased (Investigations) | 1 | 2 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Prior to publication, Investigator shall submit to the Sponsor a copy of any proposed publication. Sponsor shall have sixty (60) days to review the proposed publication for possible disclosure of Sponsor's Confidential Information and, upon request of Sponsor, Investigator shall delete any of Sponsor's Confidential Information or withhold submission of such publication to allow Sponsor to protect its intellectual property rights.